CLINICAL TRIAL: NCT05040880
Title: A Bioequivalence Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety After Administration of TELMIONE PLUS TAB. 80/12.5mg and MICARDIS PLUS TAB. 80/12.5mg in Healthy Adult Volunteers
Brief Title: A Bioequivalence Study Between Telmione Plus 80/12.5mg and Micardis Plus 80/12.5 mg in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_TMP_101
Record Dates: First submitted 2021-08-25; First posted 2021-09-10 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): TRTR
  Interventions: Drug: Telmione plus 80/12.5mg; Drug: Micardis plus 80/12.5mg
- Sequence B (Experimental): RTRT
  Interventions: Drug: Telmione plus 80/12.5mg; Drug: Micardis plus 80/12.5mg

INTERVENTIONS:
Drug: Telmione plus 80/12.5mg — Test drug (Fixed-dose combination drug of telmisartan 80mg and hydrochlorothiazide 12.5mg)
Drug: Micardis plus 80/12.5mg — Reference drug (Fixed-dose combination drug of telmisartan 80mg and hydrochlorothiazide 12.5mg)

SUMMARY:
To compare the pharmacokinetics and safety after a single dose administration of Telmione plus® 80/12.5mg and Micardis plus® 80/12.5mg in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged ≥ 19 years at screening
* Body weight ≥ 50kg and Body mass index (BMI) in the range of 18.0 and 30.0 kg/㎡
* Subjects who do not have congenital or chronic diseases requiring treatment and have no pathological symptoms or findings as a result of physical examination
* Determined by the investigator to be eligible for study participation based on the results of screening tests (clinical laboratory tests, vital signs, physical examination, 12-lead ECG) conducted according to the IP characteristics
* Subjects who decided to participate in the study and signed informed consent form voluntarily after receiving detailed explanation of the study and fully understanding

Exclusion Criteria:

* Subjects with a presence and a history of clinically significant hepatic, renal, neurology, psychiatric, pulmonary, endocrine, hematologic, oncologic, genitourinary, cardiovascular, gastrointestinal, musculoskeletal disease
* Pregnant(positive urine HCG) or breastfeeding women if female
* Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Subjects with a presence and a history of surgery or gastrointestinal diseases which might significantly change absorption of medicines
* Subjects with hypersensitivity or a history of clinically significant hyper sensitivity to ingredients with IPs, excipients, other drugs including sulfonamide and renin-angiotensin class
* Subjects with the following results in clinical laboratory tests

  * AST/ALT/ALP/γ-GTP/Bilirubin total > UNL (upper normal limit) × 2
  * Creatinine in plasma which is outside the accepted normal range or eGFR calculated by MDRD < 60 mL/min/1.73 ㎡
  * CK > UNL × 2
* Subjects with a history of drug abuse or positive to drug abuse at urine drug screening test
* Subjects with systolic blood pressure (SBP) ≥ 140 mmHg or ≤ 90 mmHg, diastolic blood pressure (DBP) ≥ 100 mmHg or ≤ 60 mmHg, or pulse rate (PR) ≤ 40 bpm or ≥ 100 bpm on vital signs measured in sitting position after taking a rest for at least 3 minutes during screening test
* Subjects with clinically significant opinions including the following results in 12-lead ECG test during screening test

  * QTc > 450 ms
  * PR interval > 200 ms
  * QRS duration > 120 ms
* Subjects who have an abnormal diet that can affect ADME of drugs or consume foods that can affect drug metabolism
* Subjects who have taken any prescription drugs or herbal medicine within 2 weeks prior to the 1st IP administration, or any over-the-counter (OTC) drug, health functional food or vitamin preparation within 10 days to the 1st IP administration (However, can participate in the study if otherwise eligible in the judgment of the investigator)
* Subjects who have taken the drug which can induce or inhibit drug metabolism enzyme within 1 month prior to the 1st IP administration
* Subjects who have participated in any other clinical study or bioequivalnece study within 6 months prior to the 1st IP administration(However, the criterion for termination of participation in other clinical study or bioequivalence study is the last administration date, and the next day is counted as one day.)
* Subjects who have donated whole blood within 2 months prior to the 1st IP administration or have donated blood components or received transfusion within 1 month prior to the 1st IP administration
* Subject who have continued drink of alcohol (> 21 units/week, 1 unit = 10 g = 12.5 mL of pure alcohol) within 6 months prior to the 1st IP administration or are unable to stop drinking from the time of signing the informed consent form to post study visit

  * alcohol (g) = intake volume(mL) × level(%) × 0.8
* Subject who have a history of excessive smoking (> 10 cigarettes/day) within 3 months prior to the 1st IP administration and unable to stop smoking from 24 hours before the administration at each period to the last sampling time at each period
* Subjects who take or are unable to stop foods containing grapefruit from 48 hours before the 1st IP administration to post study visit
* Subject who take or are unable to stop foods containing caffeine(coffee, green tea, black tee, soda, coffee-flavored milk, nutritive tonic drink) from 24 hours before the administration at each period to the last sampling time at each period
* Subjects who have exercised vigorously exceeding the level of daily life during the period from 48 hours before the 1st administration to post study visit, or who are unable to stop vigorous exercise
* Subjects or their spouse or partner who are not using an approved method of contraception or even if are not planning to become pregnant (e.g., contraceptive administration and implantation, intrauterine device, Those who are not using procedures (vasectomy, tubal ligation, etc.) from the time of written consent of the subject until two weeks after the last bioequivalence study drug administration date
* Subjects who have determined that the investigator is unsuitable to participate in the bioequivalence test due to reasons other than the above selection/exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Cmax of telmisartan | Up to 72 hours
AUClast of telmisartan | Up to 72 hours
Cmax of hydrochlorothiazide | Up to 72 hours
AUClast of hydrochlorothiazide | Up to 72 hours

SECONDARY OUTCOMES:
Tmax of telmisartan | Up to 72 hours
AUCinf of telmisartan | Up to 72 hours
t1/2 of telmisartan | Up to 72 hours
CL/F of telmisartan | Up to 72 hours
Vd/F of telmisartan | Up to 72 hours
Tmax of hydrochlorothiazide | Up to 72 hours
AUCinf of hydrochlorothiazide | Up to 72 hours
t1/2 of hydrochlorothiazide | Up to 72 hours
CL/F of hydrochlorothiazide | Up to 72 hours
Vd/F of hydrochlorothiazide | Up to 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea